CLINICAL TRIAL: NCT04495465
Title: Effects of Radial Shock Waves Therapy in the Treatment of Neck Pain: Randomized Clinical Trial
Brief Title: Effects of Radial Shock Waves Therapy in the Treatment of Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, NOELIA ZAGALAZ ANULA, Health Sciences Department Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UJAShockWavesNeck2020
Record Dates: First submitted 2020-07-27; First posted 2020-07-31 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Neck Pain; Musculoskeletal Manipulations; Extracorporeal Shockwave Therapy
Keywords: Neck Pain; Musculoskeletal Manipulations; Extracorporeal Shockwave Therapy
MeSH Terms: conditions — Neck Pain | interventions — Extracorporeal Shockwave Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Two groups: experimental group and placebo group, receiving the intervention at the same time
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: manual therapy + shock waves (Experimental): Four sessions (one per week along one month) of manual therapy (25 minutes of massage on neck muscles) and 3 minutes (2000 shocks aproximately) of extracorporeal radial shock waves therapy on painful points of neck muscles at 2 bars and 10 Hetzs.
  Interventions: Other: Radial Shock Wave Therapy; Other: Manual Therapy
- Control group: manual therapy + placebo shock waves (Placebo Comparator): Four sessions (one per week along one month) of manual therapy (25 minutes of massage on neck muscles) and 3 minutes (2000 shocks aproximately) of placebo extracorporeal radial shock waves therapy on painful points of neck muscles.
  Interventions: Other: Manual Therapy; Other: placebo shock waves

INTERVENTIONS:
Other: Radial Shock Wave Therapy — 2000 shots of extracorporeal radial shock waves therapy on neck muscles at 4bars and 10 Hertzs
  Other Names: Extracorporeal Shockwave Therapy
  Arms: Experimental group: manual therapy + shock waves
Other: Manual Therapy — 25 minute massage to neck muscles
  Other Names: Musculoskeletal Manipulations
Other: placebo shock waves — 3 minutes of placebo extracorporeal radial shock waves therapy on painful points of neck muscles.
  Arms: Control group: manual therapy + placebo shock waves

SUMMARY:
The aim of this study is to assess the effects of radial shock wave therapy in neck pain. For this objective, subjects recruited will be allocated in an experimental group or a placebo group. Both groups will receive one manual therapy and radial shock waves therapy (real for experimental group, a sham device for placebo group) session per week along one month. Neck pain, neck function, temporomandibular pain, temporomandibular function and quality of life measured will be performed before the intervention, after the last treatment and at one month follow-up.

DETAILED DESCRIPTION:
Neck pain is defined as discomfort or more intense forms of pain that are localized to the cervical region. The multifactorial etiology of neck pain includes trauma, ergonomic factors such as inappropriate postures, repetitive movements, strong physical activity, individual factors such as age, BMI, genetic factors, behavioral factors, and psychosocial factors.

The prevalence of cervicalgia ranges from 16.7 to 75.1%, of which 50% will resolve within a short time and the other half will suffer pain for a longer time. There is a higher prevalence in widows and separated, people with few economic resources, jobs that involve physical effort, low educational level, anxiety and depression. Furthermore, there is a high relationship between cervical pain and temporomandibular disorders.

From this study, the investigators are going to carry out a non-invasive, analgesic, antiinflammatory treatment and without negative side effects for the patient through radial extracorporeal shock waves (rESWT), and manual therapy (TM). Among the effects produced by shock waves the investigators find that they improve circulation due to increased blood flow and oxygenation, at tissue level the permeability of the membrane increases and its metabolic process, therefore facilitating the activation of tissue regeneration processes experiencing dystrophic changes. Furthermore, shock waves cause anti-inflammatory effects and muscle relaxation.

The main objective of the study is to evaluate the capacity of the shock waves to improve the alterations due to neck pain. To meet the above objective, a single-blind randomized clinical trial study has been designed. The selected subjects will be of legal age diagnosed with neck pain and those subjects that due to their own characteristics are not able to carry out the study will be excluded. Subjects will receive a weekly physical therapy session for four weeks. Subjects will be randomly assigned to two groups: T1 intervention group consisting of subjects who will receive manual therapy treatment and shock waves and T2 placebo group in which the subjects will receive manual therapy and placebo shock waves.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed of neck pain.

Exclusion Criteria:

* Subjects who due to their own characteristics are not able to carry out the study tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Neck pain intensity | baseline
  Numeric Pain Rating Scale to assess the intensity of the neck pain. The numeric Pain Rating Scale is a self-implemented pain intensity perception scale. In this test, all the possibilities are arranged at the same level, with 0 being the absence of pain and 10 being the maximum pain the patient is capable of imagining, organized in an increasing manner from left to right; the patient only has to mark with a cross the answer considered correct.
Neck pain intensity | at one month
  Numeric Pain Rating Scale to assess the intensity of the neck pain. The numeric Pain Rating Scale is a self-implemented pain intensity perception scale. In this test, all the possibilities are arranged at the same level, with 0 being the absence of pain and 10 being the maximum pain the patient is capable of imagining, organized in an increasing manner from left to right; the patient only has to mark with a cross the answer considered correct.
Neck pain intensity | at two months
  Numeric Pain Rating Scale to assess the intensity of the neck pain. The numeric Pain Rating Scale is a self-implemented pain intensity perception scale. In this test, all the possibilities are arranged at the same level, with 0 being the absence of pain and 10 being the maximum pain the patient is capable of imagining, organized in an increasing manner from left to right; the patient only has to mark with a cross the answer considered correct.
Neck function | baseline
  Neck Disability Index. The Neck Disability Index is a questionnaire that assesses disability produced by neck pain. It consists of ten questions with six different answers that are ordered from least to most disability, with 0 corresponding to no disability and 5 corresponding to greatest disability. The result is the sum of the answers, ranging from 0 to 50. The categorization of the final result is as follows: "no disability" if the result is between 0 and 4, "moderate disability" between 15 and 24, and "complete disability" between 35 and 50.
Neck function | at one month
  Neck Disability Index. The Neck Disability Index is a questionnaire that assesses disability produced by neck pain. It consists of ten questions with six different answers that are ordered from least to most disability, with 0 corresponding to no disability and 5 corresponding to greatest disability. The result is the sum of the answers, ranging from 0 to 50. The categorization of the final result is as follows: "no disability" if the result is between 0 and 4, "moderate disability" between 15 and 24, and "complete disability" between 35 and 50
Neck function | at two months
  Neck Disability Index. The Neck Disability Index is a questionnaire that assesses disability produced by neck pain. It consists of ten questions with six different answers that are ordered from least to most disability, with 0 corresponding to no disability and 5 corresponding to greatest disability. The result is the sum of the answers, ranging from 0 to 50. The categorization of the final result is as follows: "no disability" if the result is between 0 and 4, "moderate disability" between 15 and 24, and "complete disability" between 35 and 50

SECONDARY OUTCOMES:
temporomandibular pain intensity | baseline
  Numeric Pain Rating Scale to assess the intensity of the temporomandibular pain intensity. The numeric Pain Rating Scale is a self-implemented pain intensity perception scale. In this test, all the possibilities are arranged at the same level, with 0 being the absence of pain and 10 being the maximum pain the patient is capable of imagining, organized in an increasing manner from left to right; the patient only has to mark with a cross the answer considered correct.
temporomandibular pain intensity | at one month
  Numeric Pain Rating Scale to assess the intensity of the temporomandibular pain intensity. The numeric Pain Rating Scale is a self-implemented pain intensity perception scale. In this test, all the possibilities are arranged at the same level, with 0 being the absence of pain and 10 being the maximum pain the patient is capable of imagining, organized in an increasing manner from left to right; the patient only has to mark with a cross the answer considered correct.
temporomandibular pain intensity | at two months
  Numeric Pain Rating Scale to assess the intensity of the temporomandibular pain intensity. The numeric Pain Rating Scale is a self-implemented pain intensity perception scale. In this test, all the possibilities are arranged at the same level, with 0 being the absence of pain and 10 being the maximum pain the patient is capable of imagining, organized in an increasing manner from left to right; the patient only has to mark with a cross the answer considered correct.
Temporomandibular joint function | baseline
  using Fonseca Anamnestic Index. Its structure consists of 10 questions with a three-point scale (0=no, 5= sometimes and 10= yes), with the overall score of the test ranging from 0 to 100. The FAI evaluates the presence or absence of symptoms caused by TMDs and their severity (mild, moderate and severe).
Temporomandibular joint function | at one month
  using Fonseca Anamnestic Index. Its structure consists of 10 questions with a three-point scale (0=no, 5= sometimes and 10= yes), with the overall score of the test ranging from 0 to 100. The FAI evaluates the presence or absence of symptoms caused by TMDs and their severity (mild, moderate and severe).
Temporomandibular joint function | at two months
  using Fonseca Anamnestic Index. Its structure consists of 10 questions with a three-point scale (0=no, 5= sometimes and 10= yes), with the overall score of the test ranging from 0 to 100. The FAI evaluates the presence or absence of symptoms caused by TMDs and their severity (mild, moderate and severe).
Health Related Quality of life | baseline
  12-Item Short-Form Health Survey (SF-12): is a simple and quick questionnaire compared to its predecessor, the SF-36 that is self-administered and evaluates general quality of life from physical and emotional points of view. It consists of 12 questions that are presented with a variable number of answers. The final result of the test is obtained in a more exact way by means of a statistical processing instrument that provides the value of the physical and mental summary scores with values between 0 and 100.
Health Related Quality of life | at one month
  12-Item Short-Form Health Survey (SF-12): is a simple and quick questionnaire compared to its predecessor, the SF-36 that is self-administered and evaluates general quality of life from physical and emotional points of view. It consists of 12 questions that are presented with a variable number of answers. The final result of the test is obtained in a more exact way by means of a statistical processing instrument that provides the value of the physical and mental summary scores with values between 0 and 100.
Health Related Quality of life | at two months
  12-Item Short-Form Health Survey (SF-12): is a simple and quick questionnaire compared to its predecessor, the SF-36 that is self-administered and evaluates general quality of life from physical and emotional points of view. It consists of 12 questions that are presented with a variable number of answers. The final result of the test is obtained in a more exact way by means of a statistical processing instrument that provides the value of the physical and mental summary scores with values between 0 and 100.
Headache impact in quality of life. | baseline
  The Headache Impact Test (HIT-6) is a self-administered headache questionnaire that consists of six questions with five possible answers. The possible outcomes are "never", "rarely", "sometimes", "very often" and "always". The numerical result is the sum of the answers.
Headache impact in quality of life | at one month
  The Headache Impact Test (HIT-6) is a self-administered headache questionnaire that consists of six questions with five possible answers. The possible outcomes are "never", "rarely", "sometimes", "very often" and "always". The numerical result is the sum of the answers.
Headache impact in quality of life | at two months
  The Headache Impact Test (HIT-6) is a self-administered headache questionnaire that consists of six questions with five possible answers. The possible outcomes are "never", "rarely", "sometimes", "very often" and "always". The numerical result is the sum of the answers.
Dizziness | baseline
  Dizziness measured with Dizziness Handicap Inventory: is a self-implemented scale that identifies vertigo or lack of balance. The instrument consists of 25 questions that can be answered as yes, no or sometimes. This questionnaire identifies functional, physical and emotional problems related to balance disorders. Each dimension corresponds to different questions distributed randomly throughout the test. The functionality questions correspond to items 3, 5, 6, 7, 12, 14, 16, 19 and 24, the emotional questions correspond to items 2, 9, 10, 15, 18, 20, 21, 22 and 23, and the questions on the physical dimension correspond to items 1, 4, 8, 11, 13, 17 and 25.
Dizziness | at one month
  Dizziness measured with Dizziness Handicap Inventory: is a self-implemented scale that identifies vertigo or lack of balance. The instrument consists of 25 questions that can be answered as yes, no or sometimes. This questionnaire identifies functional, physical and emotional problems related to balance disorders. Each dimension corresponds to different questions distributed randomly throughout the test. The functionality questions correspond to items 3, 5, 6, 7, 12, 14, 16, 19 and 24, the emotional questions correspond to items 2, 9, 10, 15, 18, 20, 21, 22 and 23, and the questions on the physical dimension correspond to items 1, 4, 8, 11, 13, 17 and 25.
Dizziness | at two months
  Dizziness measured with Dizziness Handicap Inventory: is a self-implemented scale that identifies vertigo or lack of balance. The instrument consists of 25 questions that can be answered as yes, no or sometimes. This questionnaire identifies functional, physical and emotional problems related to balance disorders. Each dimension corresponds to different questions distributed randomly throughout the test. The functionality questions correspond to items 3, 5, 6, 7, 12, 14, 16, 19 and 24, the emotional questions correspond to items 2, 9, 10, 15, 18, 20, 21, 22 and 23, and the questions on the physical dimension correspond to items 1, 4, 8, 11, 13, 17 and 25.

OTHER OUTCOMES:
weight | baseline
  Record of information provided by the patient about sex, age, weight, height and body weight in kilograms (kg)
height | baseline
  height in meters (m)
body mass index | baseline
  weight and height will be combined to report body mass index in kg / m ^ 2

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Lomas-Vega, PhD, Principal Investigator — University of Jaén
Locations (1):
- Clinica Fisiomedic, Dos Hermanas, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No